CLINICAL TRIAL: NCT05468424
Title: Effect of Tablet-Based Games on Executive Functions in Older Adults With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: John Puxty (Other)
Responsible Party: Sponsor-Investigator, John Puxty, Associate Professor, Chair of Geriatric Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 6035589
Record Dates: First submitted 2022-06-29; First posted 2022-07-21 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
Keywords: video games, tablet
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FarmVille (Experimental): tablet (iPad or android) based role-playing game (FarmVille)
  Interventions: Other: tablet (iPad or android) based role-playing game
- puzzle games (Active Comparator): selection of tablet (iPad or android) based word puzzles (Word Search Ultimate and Word Cookies) and image puzzles (Flow Free and Jigsaw HD)
  Interventions: Other: tablet (iPad or android) based word puzzles and image puzzles

INTERVENTIONS:
Other: tablet (iPad or android) based role-playing game — The intervention is a tablet (iPad or android) based role-playing game called FarmVille. In FarmVille the player assumes the role of a farmer tasked with tending to crops and farm animals and using what is produced to craft goods which can be sold to expand the farm. The participant is required to play FarmVille for 5 or more hours a week for 8 weeks.
  Arms: FarmVille
Other: tablet (iPad or android) based word puzzles and image puzzles — This intervention is a selection of tablet (iPad or android) word puzzles and image puzzles. One word puzzle involves "word making" (i.e., making words from a set of random letters), and the other "word searching" (i.e., finding words on a grid of letters). One image puzzle is Flow Free, a game that requires the player to connect pairs of same coloured dots positioned on a grid ranging from 5x5 to 9x9. The other image puzzle is a jigsaw. The participant is required to play these games for 5 or more hours a week for 8 weeks.
  Arms: puzzle games

SUMMARY:
The primary objective of this study is to investigate whether a tablet-based role-playing game is more effective than tablet-based word or image puzzles at improving executive functions in older adults with mild cognitive impairment. The secondary objective of this study is to investigate whether a tablet-based role-playing game will show higher levels of engagement (measured by time played) in older adults with mild cognitive impairment than tablet-based word or image puzzles.

DETAILED DESCRIPTION:
The purpose of this study is to examine the use of tablet-based (iPad or android) video games as a means of improving executive functions in older adults with mild cognitive impairment (Petersen, Smith, Waring, et al., 1999). The worldwide rising average age of the population and increasing incidence of dementia has created an urgent need for the development of effective and engaging therapies to mitigate age- and dementia-related cognitive decline. Much evidence supports the use of cognitive therapies as a means of improving general cognition in older adults. Video games may offer benefits over traditional cognitive therapies as they are challenging and fun, provide frequent feedback which motivates and encourages user engagement, and are widely available at low cost on tablet devices. This study will be implemented as a single blinded randomized control trial structured as a 2 x 2 mixed design with one repeated factor (time: pre-training, post-training) and one between-subject factor (group: treatment, active control). Forty-two older adults with mild cognitive impairment will be randomly assigned to play either a role-playing game, or a selection of word or image puzzles, for 5 or more hours a week for a period of 8 weeks. Participants can have a study partner assist them in the study. A study partner can help the participant with using the tablet and navigating menu in the game, but cannot play the game along with the participant. Participants will be assessed pre and post training with the Cambridge Brain Sciences (www.cambridgebrainsciences.com) online battery of 12 cognitive tasks. These tasks are "based on well-established paradigms from the cognitive neuroscience literature, to measure planning, reasoning, attention, and working memory abilities" (Hampshire, Highfield, Parkin, et al., 2012, p. 1236).

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* fluent in English
* diagnosis of mild cognitive impairment
* normal or corrected hearing and vision
* can operate the touch screen on an iPad
* access to a tablet (iPad or android) for 8 weeks of the study

Exclusion Criteria:

* have started taking memory medication in the last 3 months
* have experience in any of the tablet-based games included in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
response inhibition | 8 weeks
  Double Trouble (Cambridge Brain Science, n.d., p. 3) - "A variant on the Stroop task (Stroop, 1935). Three coloured words are displayed on the screen: one at the top and two at the bottom. Participants must indicate which of two coloured words at the bottom of the screen (ignoring the colour of those words) correctly describes the colour that the word at the top of the screen is written in" (p. 3). Participants have 90 seconds to solve as many problems as possible. The task is scored on the number of correctly answered problems minus the number of incorrectly answered problems.
attention | 8 weeks
  Feature Match (Cambridge Brain Science, n.d., p. 4) - "Based on the classical feature search tasks that have been used to measure attentional processing (Treisman & Gelade, 1980). Two grids are displayed on the screen, each containing an array of abstract shapes. In half of the trials the grids differ by just one shape. Participants must indicate whether or not the grid's contents are identical. Difficulty is increased or decreased by one shape depending on whether the participant got the previous trial correct" (p. 4). Participants have 90 seconds to solve as many problems as possible. The task is scored on the sum of the difficulties of all correctly answered problems minus the sum of the difficulties of all incorrectly answered problems.
verbal short-term memory | 8 weeks
  Digit Span (Cambridge Brain Science, n.d., p. 4) - "A variant on the verbal working memory component of the WAIS-R (Weschler, 1981). A sequence of numbers will appear on the screen one after another. Once the sequence is complete, participants must repeat the sequence. Difficulty is increased or decreased by one number depending on whether the participant got the previous trial correct" (p. 4). After three errors, the task ends. The task is scored on the maximum level (e.g. the problem with the highest number of digits) that the participant successfully completed.
spatial short-term memory | 8 weeks
  Spatial Span (Cambridge Brain Science, n.d., p. 6) - "A variant on the Corsi Block Tapping Task (Corsi, 1972). Sixteen squares are displayed in a 4 x 4 grid. A sub-set of the squares flash in a random sequence at a rate of 1 flash every 900 ms. Participants must repeat the sequence by clicking on the squares in the same order in which they flashed. Difficulty is increased or decreased by one square depending on whether the participant got the previous trial correct" (p. 6). After three errors, the task ends. The task is scored on the maximum level (e.g. the problem with the highest number of targets) that the participant successfully completed.
working memory | 8 weeks
  Token Search (Cambridge Brain Science, n.d., p. 6) - "Based on a test that is used to measure strategy during search behaviours (Collins et al.,1998). Boxes are displayed in random locations. Participants must find a hidden "token" by clicking on the boxes one at a time. When the token is found, it is hidden within another box. The token will not appear within the same box twice, thus, participants must search the boxes until the token has been found once in each box. If they search the same empty box twice, or search a box in which the token has previously been found, this is an error and the trial ends. Difficulty is increased or decreased by one box depending on whether the participant got the previous trial correct" (p. 6). After three errors, the task will end. The task is scored on the maximum level (e.g. the problem with the most tokens) that the participant successfully completed.
visuospatial working memory | 8 weeks
  Monkey Ladder (Cambridge Brain Science, n.d., p. 5) - "A variant on a task from the non-human primate literature (Inoue & Matsuzawa, 2007). Sets of numbered squares are displayed on the screen at random locations. After a variable interval of time, the numbers disappear leaving just the blank squares and participants must respond by clicking the squares in ascending numerical sequence. Difficulty is increased or decreased by one numbered box depending on whether the participant got the previous trial correct" (p. 5). After three errors, the task ends. The task is scored on the maximum level (e.g. the problem with the highest number of boxes) that the participant successfully completed.
visuospatial rotations | 8 weeks
  Rotations (Cambridge Brain Science, n.d., p. 6) - "Used for measuring the ability to manipulate objects spatially in mind (Silverman et al., 2000). Two grids of coloured squared are displayed to either side of the screen with one of the grids rotated by a multiple of 90 degrees. When rotated, the grids are either identical or differ by the position of just one square. Participants must indicate whether or not the grids are identical" (p. 6). Participants have 90 seconds to solve as many problems as possible. The task is scored on the sum of the difficulties of all correctly answered problems minus the sum of the difficulties of all incorrectly answered problems.
visuospatial processing | 8 weeks
  Polygons (Cambridge Brain Science, n.d., p. 4) - "Based on the Interlocking Pentagons task (Folstein et al., 1975). A pair of overlapping polygons is displayed on one side of the screen. Participants must indicate whether a polygon displayed on the other side of the screen is identical to one of the interlocking polygons. Difficulty is increased by making the differences between the polygons more subtle or decreased by making the differences between the polygons more pronounced" (p. 4). Participants have 90 seconds to solve as many problems as possible. The task is scored on the sum of the difficulties of all correctly answered problems minus the sum of the difficulties of all incorrectly answered problems.
deductive reasoning | 8 weeks
  Odd One Out (Cambridge Brain Science, n.d., p. 3) - "Based on a sub-set of problems from the Cattell Culture Fair Intelligence Task (Cattell, 1949). Nine patterns will appear on the screen. The features that make up the patterns are colour, shape, and number and are related to each other according to a set of rules. Participants must deduce the rules that relate the object features and select the pattern that do not correspond to those rules. Difficulty is increased or decreased depending on whether the participant got the previous trial correct" (p. 3). Participants have 3 minutes to solve as many problems as possible. The task is scored on the number of correctly answered problems minus the number of incorrectly answered problems.
verbal reasoning | 8 weeks
  Grammatical (Cambridge Brain Science, n.d., p. 5) - "Based on Baddeley's three minute grammatical reasoning task (Baddeley, 1968). Short sentences describing the relationship of two shapes along with an image of the shapes are displayed on the screen. Participants must indicate whether the sentence correctly describes the pair of objects displayed on the screen" (p. 5). Participants have 90 seconds to solve as many problems as possible. The task is scored on the number of correctly answered problems minus the number of incorrectly answered problems.
planning | 8 weeks
  Spatial Planning (Cambridge Brain Science, n.d., p. 7) - "A direct descendant of the 'Tower of London' planning task (Shallice, 1982). When the task begins, numbered beads are positioned on a tree-shaped frame. Participants must reposition the beads so they are configured in ascending numerical order, in as few moves as possible. Problems become progressively harder" (p. 7). Participants have three minutes to solve as many problems as possible. The task is scored by subtracting the total number of moves made from twice the minimum number of moves required.

SECONDARY OUTCOMES:
engagement | 8 weeks
  The participants are given a Game Play Log on which they log daily the (1) minutes played, (2) minutes of study partner assistance provided, and (3) level achieved in the game.

CONTACTS AND LOCATIONS:
Overall Officials: John Puxty, MD, Principal Investigator — Providence Care Hospital; Nicole Anderson, PhD, Principal Investigator — Baycrest Academy
Locations (2):
- Canada (2):
  - Providence Care Hospital, Kingston, Ontario
  - Baycrest Academy, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baddeley, AD (1968). A 3 min reasoning test based on grammatical transformation. Psychonomic Science, 10(10), 341-342.
- [Background] Cambridge Brain Sciences (n.d.). Cambridge Brain Sciences Task Overview. Retrieved from https://www.cambridgebrainsciences.com/assets/partners/cbs-health---science-overview.pdf.
- [Background] Cattell, RB (1949). Culture free intelligence test, Scale 1, handbook.1. Institute of Personality and Ability, Champaign, Illinois.
- [Background] Collins P, Roberts AC, Dias R, Everitt BJ, Robbins TW. Perseveration and strategy in a novel spatial self-ordered sequencing task for nonhuman primates: effects of excitotoxic lesions and dopamine depletions of the prefrontal cortex. J Cogn Neurosci. 1998 May;10(3):332-54. doi: 10.1162/089892998562771. PMID 9869708
- [Background] Corsi, PM (1972). Human memory and the medial temporal region of the brain. Dissertation Abstracts International, 34(2-B), 891.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Hampshire A, Highfield RR, Parkin BL, Owen AM. Fractionating human intelligence. Neuron. 2012 Dec 20;76(6):1225-37. doi: 10.1016/j.neuron.2012.06.022. PMID 23259956
- [Background] Inoue S, Matsuzawa T. Working memory of numerals in chimpanzees. Curr Biol. 2007 Dec 4;17(23):R1004-5. doi: 10.1016/j.cub.2007.10.027. No abstract available. PMID 18054758
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Shallice T. Specific impairments of planning. Philos Trans R Soc Lond B Biol Sci. 1982 Jun 25;298(1089):199-209. doi: 10.1098/rstb.1982.0082. PMID 6125971
- [Background] Silverman I I, Choi J, Mackewn A, Fisher M, Moro J, Olshansky E. Evolved mechanisms underlying wayfinding. further studies on the hunter-gatherer theory of spatial sex differences. Evol Hum Behav. 2000 May 1;21(3):201-213. doi: 10.1016/s1090-5138(00)00036-2. PMID 10828558
- [Background] Stroop, JR (1935). Studies of interference in serial verbal reactions. Journal of Experimental Psychology, 18(6), 643-661. doi: 10.1037/h0054651.
- [Background] Treisman AM, Gelade G. A feature-integration theory of attention. Cogn Psychol. 1980 Jan;12(1):97-136. doi: 10.1016/0010-0285(80)90005-5. No abstract available. PMID 7351125
- [Background] Wechsler. D. (1981). Wechsler Adult Intelligence Scale - Revised. Manual. New York: Psychological Corporation.